CLINICAL TRIAL: NCT02580825
Title: Biofeedback Gait Retraining to Reduce Lower Extremity Impact in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MeirMc0189-15CTIL
Record Dates: First submitted 2015-09-29; First posted 2015-10-20 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2017-01

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; Ground reaction force; Knee pain
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biofeedback gait retraining (Active Comparator): The intervention program will take four weeks while in each week their will be two exercise sessions and a total of 8 sessions. Each session length is about 9 minutes. Each session will include a continuous exercise in which the patient will do walking, walking pace and running (3 minutes each section). During the meeting, participant will receive biofeedback that will displayed on a computer screen that shows the forces that develop in the knee joint so that the patient can see graphically the forces that develop around the knee joint and will be guided / try to reduce the values of the graph by changing the intensity of his landing on the tracks. In all training the time that the biofeedback is shown will be reduced.
  Interventions: Behavioral: Biofeedback gait retraining
- Exercise (Active Comparator): The control group will receive the same training program: four weeks while in each week their will be two exercise sessions and a total of 8 sessions. Each session length is about 9 minutes. Each session will include a continuous exercise in which the patient will do walking, walking pace and running (3 minutes each section). This group will not provide the biofeedback.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Biofeedback gait retraining — Each session will include a continuous exercise in which the patient will do walking, walking pace and running (3 minutes each section). During the meeting, participant will receive biofeedback that will displayed on a computer screen that shows the forces that develop in the knee joint so that the patient can see graphically the forces that develop around the knee joint and will be guided / try to reduce the values of the graph by changing the intensity of his landing on the tracks. In all training the time that the biofeedback is shown will be reduced.
  Arms: Biofeedback gait retraining
Behavioral: Exercise — Each session will include a continuous exercise in which the patient will do walking, walking pace and running (3 minutes each section).
  Arms: Exercise

SUMMARY:
The purpose of the study is to explore if self biofeedback program can reduce ground reaction force (GRF) from the lower extremity of the body and in the knee in particular and help obese children to avoid knee injuries.

DETAILED DESCRIPTION:
This study will include approximately 50 patients, aged 7-12 years. All participants and their parents will sign an informed consent form before entering the study. At the beginning, participants are asked to answer a "vas scale" questionnaire for pain. Participants will be recruited from the population of overweight children from children's sports medical center 'Meir' in Kfar Saba. In the first stage the participants will be divided randomly into two groups of intervention and control. All children will take a test of 1 km and will be instructed to walk in the maximum phase before running (at the maximum it that the child can go without running) for calculating and determine the rate of 1.0 during the assessment of the intervention program for each participant. In addition, measures of the knees (valgus) will be made by a Goniometer, which is a protractor that measures angles between bones at a precise angle.

Each participant will fill a questionnaire about pain and difficulty from which he suffers in the knee. Participants will describe to the researcher the degree of pain and / or discomfort in motion (such as walking, running) and then pass a physical examination to diagnose a knee injury.

The intervention program will take four weeks while in each week their will be two exercise session and a total of 8 sessions. Each session length is about 9 minutes. Each session will include a continuous exercise in which the patient will do walking, walking pace and running (3 minutes each section). During the meeting, participant will receive biofeedback that will displayed on a computer screen that shows the forces that develop in the knee joint so that the patient can see graphically the forces that develop around the knee joint and will be guided / try to reduce the values of the graph by changing the intensity of his landing on the tracks (be guided to land more "light", "soft" landing with a smaller noise). In all training the time that the biofeedback is shown will be reduced. The control group will receive the same training program without providing biofeedback. Each participant will perform the test with his personality shoes. At the end of the intervention program will be a statistical comparative test of the GRF that developed in the knee Relative to each child Vs his original GRF and the group averages.

ELIGIBILITY:
Inclusion Criteria:

1. Children, boys and girls, ages 7-12.
2. Children with overweight defined as BMI percentile over 85%
3. Children who are able to perform moderate physical activity.
4. Children who are able to understand and perform simple directions according to their age.

Exclusion Criteria:

1. Participant that does not wish to participate - will not be obligated to do so, and shall not participate in the study.
2. Participants with a history of chronic knee injuries
3. Participants with a background in competitive sport will not be included in the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
GRF (ground reaction force) | 8 weeks
  Reduction of ground reaction forces in three different modes of walking at an easy pace, pace and running ,measured by accelerometers (body weight).
Anthropometric measurements | 8 weeks
  Weight (Kg)
Anthropometric measurements | 8 weeks
  Height (Cm)
Anthropometric measurements | 8 weeks
  BMI ( kg/m^2)
VAS questionnaire | 8 weeks
  Visual analog score for pain (0-5)
Physicians global assessment questionnaire | 8 weeks
  To measure quality of life (0-5)

SECONDARY OUTCOMES:
Postural deviations of the knee joint | 8 weeks
  Reduction of abnormal positions of the knee such as valgus (degrees) and varus (degrees) by goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Alon Eliakim, MD, Principal Investigator — Meir Medical Center
Locations (1):
- the sports and health center for children and youth at "Meir" medical center, Kfar Saba, Israel